CLINICAL TRIAL: NCT00004201
Title: A Randomized Phase II Trial of Cisplatin or Carboplatin With Gemcitabine in Patients With Advanced Non-Small Cell Lung Cancer
Brief Title: Gemcitabine Plus Carboplatin or Cisplatin in Treating Patients With Stage IIIB, Stage IV, or Recurrent Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Herbert Irving Comprehensive Cancer Center (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000067444; CPMC-IRB-9027
Record Dates: First submitted 2000-01-21; First posted 2004-08-30 (Estimated); Last update posted 2013-02-04 (Estimated); Status verified 2007-06

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; Cisplatin; Gemcitabine

INTERVENTIONS:
Drug: carboplatin
Drug: cisplatin
Drug: gemcitabine hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Randomized phase II trial to compare the effectiveness of gemcitabine plus carboplatin with that of gemcitabine plus cisplatin in treating patients who have stage IIIB, stage IV, or recurrent non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the response rates of gemcitabine and carboplatin vs gemcitabine and cisplatin in patients with stage IIIB, IV, or recurrent non-small cell lung cancer. II. Determine the toxicity of these two regimens in this patient population. III. Determine the time to progression and one year survival of these patients on these regimens.

OUTLINE: This is a randomized study. Patients are stratified by stage of disease and gender. Patients are randomized to one of two treatment arms. Arm I: Patients receive gemcitabine IV over 30 minutes on days 1 and 8, followed by carboplatin over 60 minutes on day 1. Arm II: Patients receive gemcitabine IV over 30 minutes on days 1 and 8, followed by cisplatin IV over 60 minutes on day 1. Treatment repeats every 3 weeks for up to 8 courses in the absence of disease progression or unacceptable toxicity. Patients are followed monthly for 3 months, every two months for 6 months, and then every 3 months thereafter.

PROJECTED ACCRUAL: A total of 80 patients (40 per treatment arm) will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed stage IIIB or IV non-small cell lung cancer (NSCLC) Recurrent NSCLC treated with radiation or surgery allowed Bidimensionally measurable disease by x-ray, CT scan, MRI, or physical exam outside of irradiation field No active CNS metastases

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 70-100% Life expectancy: At least 12 weeks Hematopoietic: WBC at least 3,500/mm3 Granulocyte count greater than 1,500/mm3 Platelet count at least 100,000/mm3 Hemoglobin at least 9 g/dL Hematocrit at least 30% Hepatic: Bilirubin no greater than 2 mg/dL PT or aPTT no greater than 1.5 times upper limit of normal (ULN) AST or ALT no greater than 3 times ULN (5 times ULN if liver metastases present) Renal: Creatinine no greater than 2 mg/dL Other: Not pregnant or nursing Fertile patients must use effective contraception during and for 3 months after study No serious concurrent systemic disorder that would preclude study compliance No active infection No second primary malignancy within the past 5 years, except: Adequately treated basal cell skin cancer Carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 3 weeks since prior biologic therapy No concurrent immunotherapy Chemotherapy: No prior chemotherapy No other concurrent chemotherapy Endocrine therapy: At least 3 weeks since prior endocrine therapy No concurrent hormonal therapy (except contraceptives and replacement steroids) Radiotherapy: See Disease Characteristics At least 3 weeks since prior radiotherapy No concurrent radiotherapy Surgery: See Disease Characteristics Other: At least 4 weeks since other prior investigational drugs No other concurrent experimental drugs No concurrent interleukin-11 for patients with cardiac disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Study Completion 2004-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Haralambos Raftopoulos, MD, Study Chair — Herbert Irving Comprehensive Cancer Center